CLINICAL TRIAL: NCT04419597
Title: Randomized Multicenter Controlled Study to Evaluate the Safety and Efficacy of HEMOPATCH® Compared to Routine Care for Dural Closure as Reinforcement for the Prevention of Postoperative Cerebrospinal Fluid Leakage (CSF) in Patients Undergoing Posterior Fossa Surgery
Brief Title: Hemopatch Safety and Efficacy Evaluation Versus Standard Practice for Sealing the Dura in Cerebrospinal Fluid Leaks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEUROHEMOPATCH
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Surgery
Keywords: Posterior fossa; HEMOPATCH; cerebrospinal fluid (CSF); CSF leak
MeSH Terms: conditions — Cerebrospinal Fluid Otorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEMOPATCH Collagen Patch and PEG Haemostatic Sealant (Experimental): Two units of the large patch are applied as reinforcement of the primary dural seal (HEMOPATCH 4,5x9cm, 1506253).
  Interventions: Device: HEMOPATCH
- Standard of care treatment (Active Comparator): Usual clinical practice techniques for reinforcing primary dural closure.
  Interventions: Device: Standard of care

INTERVENTIONS:
Device: HEMOPATCH — The treatment will be performed with the HEMOPATCH collagen patch and hemostatic PEG sealant (Baxter), applying two units of the large patch to reinforce the primary dural closure (HEMOPATCH 4.5x9cm, 1506253).
  Arms: HEMOPATCH Collagen Patch and PEG Haemostatic Sealant
Device: Standard of care — Usual clinical practice techniques for reinforcing primary dural closure.
  Arms: Standard of care treatment

SUMMARY:
Posterior fossa surgeries are generally complicated by difficulties in creating a watertight dural closure, which often requires the use of dural substitutes. In particular, surgical procedures at this location are associated with an increased rate of fluid leakage (cerebrospinal fluid (CSF)) or inflow (blood, air, etc.) creating hydrodynamic complications. Effective sealing of the dura is required to prevent such complications and infections by minimizing the introduction of irritating blood products into the CSF. Since true hermetic dural seals are often impossible to achieve, dural sealants have been developed that can be applied to the sutured dural perimeter to help prevent complications related to CSF. Adjuvant use of such sealants may be prudent, particularly in posterior fossa surgeries, as the incidence of CSF leakage has been reported to be as high as approximately 15-28% with such surgeries, with an increased risk of leakage. 5.84 times greater than supratentorial procedures.

DETAILED DESCRIPTION:
Various techniques have been developed to overcome this problem and achieve a tight dural closure. Although there is published evidence showing the efficacy and safety of some of these sealants in posterior fossa surgery, the different types of pathologies and various population risk factors included in these trials make it difficult to interpret the results. Having selective inclusion criteria and including patients with a selected pathology could be essential to obtain clearer results.

Postoperative CSF leak has two aspects: one is pseudomeningocele (a subcutaneous collection of CSF); the other is a CSF fistula in which CSF reaches the skin. This second one is much more dangerous and constitutes one of the most important complications of this surgery, but the pseudomeningocele is a clinical demonstration of failure of the dural closure.

HEMOPATCH is a soft, thin, foldable and flexible collagen patch, coated with NHS-PEG. HEMOPATCH is indicated as a hemostatic device and surgical seal for procedures in which control of bleeding or leakage of other body fluids or air by conventional surgical techniques is ineffective or impractical.

Preliminary clinical evidence collects a prospective case series of 200 patients, in which the authors reviewed the use of HEMOPATCH for dural augmentation in high-risk patients from 2014 to this year. After 2 years of refining the technique, a decrease in CSF leaks from 27% to 7% was achieved, and no adverse events related to the application of the product were observed. A retrospective cohort study has recently been published comparing the use of HEMOPATCH versus routine clinical practice in 290 patients, in which 147 used standard dural reinforcement techniques, and 143 used HEMOPATCH. The CSF fistula appearance rates were 7.69% in the HEMOPATCH group, compared to 32.65% in the control group.

These recent results, along with the characteristics and properties of the patch, could make this sealant a safe and plausible option to achieve sealing after posterior fossa surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned for non-traumatic posterior fossa surgery
* Surgery that requires opening and closing of the dura mater.
* Patients who have a clean surgical wound (class I surgical wound classification)
* Patients undergoing one of the following surgical procedures:
* Space occupant injuries (LOEs) rese dried through the following approaches:
* Approaching the rear pit of the middle line
* Approach to the posterior paramedian fossa
* Approach to the cerebellar pontine angle (PC) and the back of the petrous vertex
* Clinical diagnosis of primary Chiari 1 (CM1) malformation and scheduled decompression surgery, with evidence of NM of tonsil herniation down by an independent official radiology report.
* Subjects who are able to provide written informed consent prior to participating in the clinical trial.
* Be over 18 years of age.
* Understand the purpose of the study and be available for frequent hospital visits.
* Women of childbearing potential and males with partners of childbearing potential should commit to using a highly effective method of contraception (such as surgical sterilization, double barrier method, oral contraceptives or contraceptive hormonal implants) and to continue to use them for up to 6 months after surgery.

Exclusion Criteria:

* Patients undergoing a supratentorial surgical procedure/approach.
* Patients undergoing any other approach/surgical procedure at the base of the skull that is not in the posterior pit:
* Side boarding of the foramen magno: far side, extreme side, anterolateral, posterolateral,
* Approaching the jugular foramen: infratemporal, condylar juxta, transjugular
* Approach to the middle pit: subtemporal (+/-petrous apex perforation), pterional approach (any temporary fronto approach +/- orbitozygomatic replacement)
* Approach to the previous pit: subfrontal (uni or bilateral)
* Presence of hydrocephalus not resolved prior to surgery
* Previous surgery in the posterior pit.
* Pre-radiation therapy treatment.
* Previous (within the last 6 months) or anticipated neurosurgical procedure involving the opening of the dura mater that may affect the safety assessment
* > 1 dural opening
* Inability to understand informed consent or unwillingness to participate in the study.
* Inability, at the time of consent, to return for follow-up evaluations after surgery
* Evidence of spinal dysraphism.
* Allergy, hypersensitivity or history of allergic reaction to Hemopatch or its components (to bovine proteins or bright blue dye: FD&C blue No. 1 [blue 1]).
* Evidence of an infection within 5 days prior to the start of the study.
* Pregnancy or planning to become pregnant during the course of the study. Breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
proportion of participants with clinically evident CSF leak after the operation up to 4 weeks. | 4 weeks
  Clinically evident CSF leak, observed from the operation to 4 weeks later. It will be measured every 24 hours until the patient is discharged. The following measurement will be made at the visit of the 4 weeks (+/- 7 days) from the operation

SECONDARY OUTCOMES:
Proportion of participants with clinical pseudomeningocele or evident MRI | 6 months
  Clinical evidence of Pseudomeningocele or by imaging techniques, evaluated by CT or MRI during the 4 postoperative weeks, by MRI at 6 postoperative months, or at any visit of patients within 6 postoperative months according to the criteria of the investigator
Proportion of participants with ascent of the cerebellar tonsils | 6 months
  The elevation of the cerebellar tonsils will be measured, according to the baseline preoperative CT / MRI, in the MRI test performed 6 months after the operation.
Proportion of participants with readmissions related to CSF leaks | 4 weeks
  The need for readmission / reoperation related to CSF leak will be collected up to 4 weeks after the operation.
Number of Participants with Surgical site infections (SSI) | 4 weeks
  Bacterial or chemical meningitis (SSI)
Assessment of quality of life (QoL): SF12 questionnaire (Short Form 12 questionnaire) | 6 months
  The SF-12 measures overall quality of life and includes items that assess participation. The SF-12 is a frequently used measure and has shown to have good internal consistency, reliability, construct validity and responsiveness in patients with chronic (low) back pain (Luo et al., 2003). The measure is a subset of 12 items from the SF-36 including 6 items from the physical summary measure (PCS) and 6 items from the mental summary measure (MCS).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No